CLINICAL TRIAL: NCT05114889
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 1 Clinical Trial to Evaluate Safety and Tolerability of BSI-045B mAb Injection in Healthy Adult Subjects and Patients With Atopic Dermatitis
Brief Title: Safety and Tolerability of BSI-045B in Healthy Adult Subjects and Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosion, Inc. (Industry)
Collaborators: Southern Star Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BSI-045B-001
Record Dates: First submitted 2021-09-09; First posted 2021-11-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Ascending Dose Healthy Volunteer (Experimental): BSI-045B
  Interventions: Biological: BSI-045B
- Multiple Ascending Dose Healthy Volunteer (Experimental): BSI-045B
  Interventions: Biological: BSI-045B
- Single Dose Atopic Dermatitis patients (Experimental): BSI-045B
  Interventions: Biological: BSI-045B

INTERVENTIONS:
Biological: BSI-045B — BSI-045B will be administered weekly, subcutaneously

SUMMARY:
This randomized, double-blind, single center, placebo-controlled, phase 1 single ascending dose (SAD)/multiple ascending dose (MAD) study is designed to assess the safety, tolerability, PK, activity, immunogenicity, and PD of BSI-045B. Approximately 68 subjects will be enrolled. Subjects in this study include 56 healthy volunteers (HVs) and 12 patients with AD.

This study is divided into 3 parts:

1. Part A: Evaluate the safety, tolerability, PK, immunogenicity, and PD of single ascending doses of BSI-045B administered as a subcutaneous (SC) injection of 120, 240, 480, and 720 mg to HVs
2. Part B: Evaluate the safety, tolerability, PK, activity (as measured by the Eczema Area and Severity Index [EASI] score), immunogenicity, and PD of a single dose of BSI-045B administered as a SC injection of 480 mg to patients with AD
3. Part C: Evaluate the safety, tolerability, PK, immunogenicity, and PD of multiple ascending doses of BSI-045B administered as five (5) SC injections of 240, 480, and 600 mg every 7 days (Q7D) to HVs

DETAILED DESCRIPTION:
This study is a phase 1 clinical study to evaluate the safety, tolerability, immunogenicity, PK profile, activity, and PD of BSI-045B injection after single/multiple doses in adult HVs and patients with AD using a randomized, double-blind, placebo-controlled design. It consists of 3 parts: a SAD study in HVs, a single dose study in patients with AD, and a MAD study in HVs.

Part A: Single Ascending Dose in HVs The SAD study in HVs will consist of single ascending doses in a 4-cohort design. Cohorts 1, 2, 3, and 4 will each consist of 8 HVs (6 Active: 2 Placebo). The total number of HVs to be enrolled in Part A is 32.

Subjects in Part A will be enrolled as follows:

Cohort 1: HVs (Active:Placebo 6:2), 120 mg, single dose; n = 8 Cohort 2: HVs (Active:Placebo 6:2), 240 mg, single dose; n = 8 Cohort 3: HVs (Active:Placebo 6:2), 480 mg, single dose; n = 8 Cohort 4: HVs (Active:Placebo 6:2), 720 mg, single dose; n = 8 The preferred SC injection site is the abdomen. Multiple SC injections required for higher dose cohorts should be administered no more than 1 minute apart. The thigh can be used as an alternative site for SC injections. In Cohort 1, a 1 mL injection of 120 mg/mL (120 mg total dose) will be administered at a single SC injection site. In Cohort 2, a 2 mL injection of 120 mg/mL (240 mg total dose) will be administered at a single SC injection site. In Cohort 3, two 2 mL injections of 120 mg/mL will be administered simultaneously at 2 separate SC injection sites for a total of 4 mL (480 mg total dose). In Cohort 4, three 2 mL injections of 120 mg/mL will be administered simultaneously at three separate SC injection sites, for a total of 6 mL (720 mg total dose).

Part B: Single Dose in Patients with AD The total number of patients with AD to be enrolled in the single-dose study in Part B is 12.

Following a thorough assessment of safety, tolerability, and PK at Week 11 and Week 12 of the HVs treated with 480 mg in Part A, subjects will be enrolled into Part B (so that Day 1 of Part B will correspond to Day 1 of Week 13 of Part A).

Patients with AD will be enrolled as follows:

Cohort 1: Patients with AD (Active:Placebo 9:3), 480 mg, single dose; n = 12 The preferred SC injection site is the abdomen. Injections should be administered no more than 1 minute apart. The thigh can be used as an alternative site for SC injections. Patients with AD will be administered two separate 2 mL injections of 120 mg/mL simultaneously at two separate SC injection sites, for a total of 4 mL (480 mg total dose).

Management of SAD HV Cohort (Part A) and Single-Dose Cohort, Patients with AD (Part B) Healthy volunteers and patients with AD will be admitted to the phase 1 clinical site 1 day before each dose administration. In this phase 1 study of BSI-045B, sentinel dosing will be used for each of the SAD cohorts. The first 2 HVs and AD patients in each cohort will receive either BSI-045B or placebo in parallel (1 Active:1 Placebo), followed by a 3 day gap to allow for the evaluation of safety and tolerability before administering the same dose of BSI-045B or placebo to the remaining HVs (5 Active:1 Placebo) or AD patients (8 Active:2 Placebo).

Healthy volunteers and patients with AD will be confined at the clinical site to assess tolerability, safety, and adverse events (AEs), and for collection of blood samples for PK analysis. After 9 days of evaluation, HVs or patients with AD will leave the phase 1 clinic after completion of the clinical assessments. Follow-up visits at scheduled time points will be conducted to evaluate safety, tolerability, PK, immunogenicity, and biomarkers.

All decisions concerning dose escalation will be made by a Safety Review Committee composed of representatives from Biosion (at a minimum, the clinical science representative and pharmacovigilance physician, or appropriate delegates), the Principal Investigator and an independent member. The Investigator, Biosion personnel, and HVs or patients will remain blinded throughout the study. Pharmacy staff preparing the study medications will be unblinded. If unblinding is necessary for a specific subject, emergency unblinding may be arranged after approved by the Principal Investigator and discussed with the Medical Monitor. Dose escalation meetings will be carried out in accordance with the Safety Review Committee Charter.

Follow-up assessments will occur on Day 15 and during subsequent visits to the clinic for PK blood draws through Day 113 (the termination of each cohort in the SAD study). Adverse events will be collected through Day 113 to determine whether there are ongoing AEs, serious adverse events (SAEs), worsening of AEs or SAEs, or development of new AEs or SAEs. Concomitant medications taken after the final dose of BSI-045B or placebo will be recorded through Day 113. Follow-up will occur during clinic visits and if abnormal, clinically significant findings are observed upon discharge. At the Investigator's discretion, volunteers may be brought back to the clinic for re-evaluation.

Part C: Multiple Ascending Doses in HVs The MAD study will consist of multiple ascending doses in 3 cohorts. Cohorts 1, 2, and 3 will consist of 8 HVs (6 Active:2 Placebo). The MAD study will enroll a total of 24 HVs.

The MAD Part C portion of the study will commence after pharmacokinetic and safety information from the 2nd cohort (240 mg total dose) of the HV SAD portion of the study has been evaluated and approved by the Safety Review Committee. Sequential groups of HVs will receive SC injections of BSI-045B Q7D for a total of 5 doses. BSI-045B (or placebo) will be administered as single- or multiple-site SC injection(s).

Subjects in Part C will be enrolled as follows:

Cohort 1: HVs (Active:Placebo 6:2), 240 mg Q7D, 5 doses; n = 8 Cohort 2: HVs (Active:Placebo 6:2), 480 mg Q7D, 5 doses; n = 8 Cohort 3: HVs (Active:Placebo 6:2), 600 mg Q7D, 5 doses; n = 8 Healthy volunteers will be admitted to the phase 1 clinical site 1 day before each dose administration and will be discharged on Day 9 (after dose 2 on Day 8), the following day, 24 h post-dose for doses 3 and 4 and on Day 37 after dose 5. BSI-045B or placebo will be administered in the morning of the first day of each administration. The preferred SC injection site is the abdomen. Multiple SC injections required for higher dose cohorts should be administered no more than 1 minute apart. The thigh can be used as an alternative site for SC injections. For each dose administration, SC dosing should alternate between the left and right sides of the abdomen or left and right thigh. In Cohort 1 (240 mg), a 2 mL injection of 120 mg/mL will be administered at a single SC injection site. For Cohort 2 (480 mg), two 2 mL injections of 120 mg/mL of drug or placebo will be administered simultaneously at two separate SC injection sites, for a total of 4 mL. In Cohort 3 (600 mg), two separate 2 mL injections of 120 mg/mL of drug or placebo and a 1 mL injection of 120 mg/mL will be administered simultaneously at 3 separate SC injection sites, for a total of 5 mL.

Healthy volunteers will be confined to the clinic to assess safety, tolerability, PK, and immunogenicity. Adverse events will be recorded and blood samples will be collected for PK analysis. After 9 days of evaluation, HVs will leave the phase 1 clinic after the PK blood draw. Follow-up visits will be conducted at scheduled time points. HVs will return for admission to the unit 1 day prior to dosing for doses 3, 4 and 5 on Days 15, 22, and 29 respectively, and will be discharged 24 h post dose after doses 3 and 4 and on Day 37 after the final dose (dose 5).

ELIGIBILITY:
Inclusion Criteria:

* Subject eligibility is determined according to the following criteria prior to entry into the study:

  1. In the opinion of the Investigator, the subject is capable of understanding and complying with protocol requirements.
  2. The subject signs and dates a written Informed Consent Form (ICF) and any required privacy authorization prior to the initiation of any study procedures.
  3. The subject is a healthy adult male or female.
  4. The subject is aged 18 to 55 years, inclusive at the time of consent.
  5. A female subject weighs at least 45 kg and a male subject weighs at least 50 kg. The subject has a body mass index (BMI) between 18.0 and 32.0 kg/m2 inclusive at Screening.
  6. A male subject who is non-sterilized and sexually active with a female partner of childbearing potential agrees to use highly effective contraception from the time of signing the ICF throughout the duration of the study and for 90 days (~5 half-lives) have elapsed since the last dose of study drug. Examples of highly effective contraception can be found in Appendix 1.
  7. A female subject of childbearing potential who is sexually active with a non-sterilized male partner agrees to routinely use highly effective contraception from the time of signing the ICF throughout the duration of the study and for 90 days have elapsed since the last dose of study drug. Examples of highly effective contraception can be found in Appendix 1.
  8. The subject has a negative urine/blood result for drugs of abuse (defined as any illicit drug use) at Screening or on Day -1.

Exclusion Criteria:

* Any subject who meets any of the following criteria will not qualify for entry into the study:

  1. The subject has received any investigational compound within 30 days or five half-lives (whichever is greater) prior to the first dose of study drug.
  2. The subject is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of the study (e.g., spouse, parent, child, sibling) or makes consent under duress.
  3. The subject has any clinically significant illness, such as cardiovascular, neurologic, pulmonary, hepatic, renal, metabolic, gastrointestinal, neurologic, immunologic, endocrine, or psychiatric disease or disorder, current infection with coronavirus disease 2019 (COVID-19), or other abnormality that may affect safety, increase the risk for seizure or lower the seizure threshold, or potentially confound the study results. It is the responsibility of the Investigator to assess the clinical significance of a subject's condition; however, consultation with the Biosion Medical Monitor may be warranted.
  4. The subject has a known hypersensitivity to any component of the formulation of BSI-045B.
  5. The subject has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to Screening or is unwilling to agree to abstain from alcohol and drugs throughout the study.
  6. The subject has taken any prohibited concomitant medications (Section 5.5).
  7. The subject had a major elective surgical procedure within 8 weeks prior to Day 1.
  8. The subject is pregnant or lactating or intends to become pregnant or donate ova before, during, or within 90 days (~ 5 half-lives) since the last dose of study drug.
  9. If male, the subject intends to donate sperm during the course of this study or within 90 days (~ 5 half-lives) since the last dose of study drug
  10. The subject has had previous episodes of seizures or convulsions (lifetime) including absence seizure and febrile convulsion.
  11. The subject or any immediate family member has a history of epilepsy (including febrile convulsions).
  12. The subject has a history of neurologic abnormalities including abnormal electroencephalography, brain injury including traumatic injury, perinatal cerebropathy, postnatal brain damage, blood-brain barrier abnormality, and cavernous angioma.
  13. The subject has a history of cerebral arteriosclerosis.
  14. The subject has a history of cancer. Subjects with basal cell carcinoma, localized squamous cell carcinoma of the skin, or carcinoma in situ of the cervix may be included in the study if they have completed curative treatment at least 12 months before the first visit. Subjects with other malignant tumors may be included if they have completed curative treatment at least 5 years before the first visit (Day 1).
  15. The subject has a positive test result for hepatitis B surface antigen (HbsAg), anti- hepatitis C virus (HCV), or a known history of human immunodeficiency virus (HIV) infection at Screening.
  16. The subject has poor peripheral venous access.
  17. The subject has donated or lost ≥450 mL of his or her blood (including plasmapheresis) or had a transfusion of any blood product within 90 days prior to Day 1.
  18. The subject has an abnormal (clinically significant) electrocardiogram (ECG) at Screening or on Day -1. Entry of any subject with an abnormal (not clinically significant) ECG must be approved and documented by signature of the Principal Investigator or medically qualified Sub-Investigator. In the case of a corrected QT interval (Fridericia) (QTcF) >450 ms or >470 ms (HVs or AD patients with bundle branch block) or PR interval outside the range of 115 to 220 ms, assessment may be repeated once for eligibility determination at Screening and/or on Day -1.
  19. The subject has a supine systolic blood pressure <90 or >144 mm Hg or a supine diastolic blood pressure <50 or >94 mm Hg. If out of range, assessment may be repeated once for eligibility determination at Screening and/or on Day -1.
  20. The subject has a resting heart rate <40 or >90 bpm (not on ECGs) and considered clinically significant by the Investigator. If out of range, the assessment may be repeated once for eligibility determination at Screening and/or on Day -1.
  21. The subject has abnormal laboratory values at Screening that suggest a clinically significant underlying disease, or the subject has the following laboratory abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 times the upper limit of normal unless otherwise agreed to by the Sponsor and Principal Investigator.

In addition to the general criteria above, AD patients in Part B must meet the following inclusion criteria to enter the study:

1. The patient has a diagnosis of AD (according to the criteria established by Hanifin et al, 2001 and Rajka et al, 1989).
2. The EASI score is ≥15 at Screening.
3. The score on the Investigator's Global Assessment is ≥3 at Screening.
4. The score on the SCORing Atopic Dermatitis instrument is ≥20 at Screening.
5. The total body surface area affected by AD is ≥10% as assessed by the EASI at Screening.
6. The patient has an inadequate response to topical medications, or topical treatment is medically inadvisable.

In addition to the general criteria above, AD patients in Part B must not meet any of the following exclusion criteria:

1. The patient has another dermatologic condition that might confound a diagnosis of AD or a treatment assessment.
2. The patient has a history of anaphylaxis following biologic therapy.
3. The patient has a history of clinically significant infections within 4 weeks prior to Day -1.
4. The patient has a diagnosis of helminthic parasitic infection within 6 months prior to Screening.
5. The patient has received any marketed or investigational biologic agent within 5 half-lives prior to Screening.
6. The patient has received treatment with immunosuppressive or immunomodulatory drugs without adequate washout, or has received phototherapy for AD within 4 weeks prior to Day 1. For drugs, an adequate washout period is 5 half-lives (e.g., 10 weeks for dupilumab).
7. The patient has initiated treatment with topical corticosteroids (TCS) or topical calcineurin inhibitors within 1 week prior to Day -1. If rescue medications are deemed warranted by the PI class IV TCS may be used as rescue medication after Day -1 (see Table 13).
8. The patient has initiated treatment with prescription moisturizers or moisturizers containing additives such as ceramide, hyaluronic acid, urea, or filaggrin degradation products during the Screening period (patients may continue to use stable doses of such moisturizers if initiated before the Screening visit, but should not change to a different product during the study).
9. The patient plans to use any other prohibited medication or undergo any prohibited procedure during the study. Oral antibiotics are permitted. Bleach baths are not permitted.
10. The patient has received any investigational compound within 30 days or 5 half-lives (whichever is greater) days prior to Day 1.
11. The subject has a risk of suicide per the Columbia-Suicide Severity Rating Scale (a score of 4 or above on ideation or any suicidal behavior) or according to the Investigator's clinical judgment, has made a suicide attempt in the previous 6 months, or has a history of deliberate self-harm in the past 6 months. A subject with a lower score may be enrolled in the study.
12. The patient has any clinically relevant abnormal finding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | baseline to 17 weeks
  The incidence of TEAEs (AEs and SAEs) summarized by system organ class and preferred term.
Laboratory Tests | baseline to 17 weeks
  Number of subjects with clinically significant change from baseline in safety lab (e.g. hematology, chemistry)
Vital signs | baseline to 17 weeks
  Number of subjects with clinically significant change from baseline in vital signs (heart rate, blood pressure, and weight)
ECG | baseline to 17 weeks
  Number of subjects with clinically significant change from baseline in ECG (rhythm, QT interval)

SECONDARY OUTCOMES:
Pharmacokinetic parameters | baseline to 17 weeks
  Such as Peak Plasma Concentration (Cmax)
Pharmacodynamics (PD) | baseline to 17 weeks
  such as change in IL-4
Immunogenicity | baseline to 17 weeks
  The number of subjects with treatment emergent anti-drug antibody (ADA)
Clinical activity | baseline to 16 weeks
  Percent of patients with 50% and 75% improvement in the Eczema Area and Severity Index (EASI) scores

CONTACTS AND LOCATIONS:
Overall Officials: Argent Christopher, Principal Investigator — Scientia Clinical Research Ltd
Locations (1):
- Scientia Clinical Research, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No